CLINICAL TRIAL: NCT03010540
Title: Emergence Delirium and Recovery Profile in Patients Undergoing Cleft Lip and Palate Repair: Comparison of Combination of Morphine and Fentanyl With Fentanyl Alone
Brief Title: Effect Of Combination of Morphine+Fentanyl on Emergence Delirium in Patients of Cleft Lip and Palate Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, DR PARUL GUPTA, Junior Resident, department of Anaesthesia and Intensive Care, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Emergence delirium
Record Dates: First submitted 2016-12-22; First posted 2017-01-05 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Anesthesia Emergence Delirium
MeSH Terms: conditions — Emergence Delirium | interventions — Morphine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Morphine Plus Fentanyl (Experimental)
  Interventions: Drug: MORPHINE PLUS FENTANYL
- Fentanyl only (Active Comparator)
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: MORPHINE PLUS FENTANYL — Effect Of Morphine Plus Fentanyl On Emergence Delirium
  Arms: Morphine Plus Fentanyl
Drug: Fentanyl — Effect Of Fentanyl Only On Emergence Delirium
  Arms: Fentanyl only

SUMMARY:
Emergence Delirium And Recovery Profile In Patients Undergoing Cleft Lip And Cleft Palate Repair With Either Combination Of Morphine Plus Fentanyl Or Fentanyl Alone

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 Patients Undergoing Cleft Lip And Palate Repair

Exclusion Criteria:

* CNS Disorders
* Respiratory Infection
* GERD

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2015-07; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Emergence Delirium ( PAED Scale) | 30 Minutes Postoperatively

SECONDARY OUTCOMES:
Post Operative Pain (FLACC Scale ) | 30 Minutes Postoperatively
Saturation Of Oxygen (SpO2 in %) | 30 Minutes Postoperatively
Temperature (degree Celsius) | 30 Minutes Postoperatively
Heart Rate (Beats Per Minute) | 30 Minutes Postoperatively
Respiratory Rate (Per Minute) | 30 Minutes Postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- PGIMER, Chandigarh, Punjab, India

IPD SHARING:
Plan to Share IPD: No